CLINICAL TRIAL: NCT00983580
Title: Randomized Phase II Trial of Aspirin and Difluoromethylornithine (DFMO) in Patients at High Risk of Colorectal Cancer
Brief Title: Acetylsalicylic Acid and Eflornithine in Treating Patients at High Risk for Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-01192; NCI-2009-01192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-001758; MC054A (Other: Mayo Clinic); R01CA113681 (NIH); P30CA015083 (NIH); NCT01647126 (obsolete NCT alias)
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Adenomatous Polyp
MeSH Terms: conditions — Adenomatous Polyps | interventions — Aspirin; Eflornithine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (acetylsalicylic acid and eflornithine) (Experimental): Patients receive acetylsalicylic acid PO once daily and eflornithine PO twice daily on days 1-28.
  Interventions: Drug: Aspirin; Drug: Eflornithine; Other: Laboratory Biomarker Analysis; Other: Telephone-Based Intervention
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO three times daily on days 1-28.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo; Other: Telephone-Based Intervention

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm I (acetylsalicylic acid and eflornithine)
Drug: Eflornithine — Given PO
  Other Names: Alpha-Difluoromethylornithine; DFMO; difluoromethylornithine; Difluromethylornithine
  Arms: Arm I (acetylsalicylic acid and eflornithine)
Other: Laboratory Biomarker Analysis — Correlative study
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Telephone-Based Intervention — Ancillary studies

SUMMARY:
This phase II trial is studying how well giving acetylsalicylic acid together with eflornithine works in treating patients at high risk for colorectal cancer. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of acetylsalicylic acid and eflornithine may prevent colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The proportion of subjects with an adenoma recurrence at the 1-year follow-up colonoscopy exam. This adenoma recurrence rate for difluoromethylornithine (DFMO) (eflornithine) + aspirin will be compared to double placebo to see if there is improvement in the adenoma recurrence rate in this patient population.

SECONDARY OBJECTIVES:

I. To determine the relative tolerability and safety of the treatment regimens administered for 12 months.

II. To determine the effect of the study drugs (aspirin [acetylsalicylic acid] + DFMO) and placebo with respect to proliferation (Ki67 labeling index), apoptosis (caspase-3 expression assay), and drug effect markers (COX-1, -2, polyamines, PGE2) from adenomas, aberrant crypt focus (ACF) and normal-appearing mucosa using pre- and 12-month post-intervention tissue biopsy samples.

III. To estimate the percentage change in rectal ACF number, as determined by magnifying colonoscopy in subjects treated for 12 months with placebo or study drugs (aspirin +DFMO) by comparing % change in drug versus placebo arms.

IV. To characterize ACF based on three criteria (ACF size [crypt number < 50 or >= 50], crypt morphology characteristics, and histology) of ACF and to correlate such characteristics with the intervention (vs placebo). Also, to evaluate the natural history of ACF over 1-year on placebo.

V. To correlate the 12-month measurements of ACF size (# crypts/ACF), number, morphology, and histopathology with the adenoma recurrence data at 12 and 36 months; correlate the 12-month % (and actual) change in ACF size and number with the 12- and 36-month adenoma recurrence rate; and correlate the adenoma recurrence data at 1 year with the adenoma recurrence data at 3 years.

TERTIARY OBJECTIVES:

I. To explore the effects of the study agents on a focused panel of tissue biomarkers in pre- and post-intervention biopsy samples from recurrent adenomas, rectal ACF, and adjacent normal-appearing mucosa among subjects enrolled in the phase II clinical trial.

II. To determine if cleaved capase-3 expression can improve the detection of apoptotic cells by recognizing cellular commitment to apoptosis prior to late nuclear morphologic features and correlate with apoptotic regulatory proteins, histology, and treatment response.

III. To determine the effects of aspirin on its biochemical targets COX-1, -2, and prostaglandin E2, and polyamine levels in subjects receiving DFMO.

IV. To examine COX-2-dependent genes (i.e., Bcl-2 and DR5) in adenomas and ACF that have been shown to regulate the intrinsic mitochondrial and extrinsic death receptor-mediated apoptotic pathways in vitro and in vivo.

V. To perform expression profiling of adenomas or ACF and to relate such date to ACF histology, size/morphology, modulation by chemopreventive agents, and subsequent adenoma recurrence rates.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive acetylsalicylic acid orally (PO) once daily and eflornithine PO twice daily on days 1-28.

ARM II: Patients receive placebo PO three times daily on days 1-28.

Treatment repeats every 28 days for 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6, 12, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior advanced adenomas
* Advanced adenomas are defined as subject with polyps >= 1 cm, tubulovillous adenomas (25-75 percent villous features), villous adenomas (> 75 percent villous), or high-grade dysplasia
* Prior colon cancer (>= 3 years out from invasive cancer)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to under and the willingness to sign a written informed consent document
* Willingness to provide mandatory tissue for research purposes
* Negative pregnancy test =< 7 days prior to randomization
* Hemoglobin (Hgb) within normal limits for institution/lab
* Platelet count >= 100,000/ul
* White blood cell count (WBC) >= 3,000/ul
* Alanine aminotransferase (ALT) =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2 x institutional ULN
* Total bilirubin =< 1.5 x institutional ULN
* Serum calcium =< institutional ULN
* Serum creatinine =< 1.5 x institutional ULN
* Colonoscopy =< 45 days prior to randomization with removal of all adenomas or polyps >= 2 mm in size

Exclusion Criteria:

* Any history of current or prior rectal cancer
* Known diagnosis of colon heritable cancer syndrome (familial adenomatous polyposis [FAP], hereditary nonpolyposis colorectal cancer [HNPCC]) or inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* Inability to swallow pills
* Bleeding diathesis
* New diagnosis of carcinoma
* History of hypersensitivity to COX-2 inhibitors, sulfonamides, nonsteroidal antiinflammatory drugs (NSAIDs), salicylates, or ursodeoxycholic acid
* History of gastroduodenal ulcers documented =< 1 year
* Known inability to participate in the scheduled follow-up tests
* Significant medical or psychiatric problems which would make the subject a poor protocol candidate, in the opinion of the treating physician
* Total colectomy
* Patients with a colostomy
* History of pelvic or rectal radiation therapy
* History of invasive carcinoma =< 5 years (except subjects with Dukes A/B1 carcinoma =< 5 years prior to pre-registration or any stage of colon cancer if >= 3 years post surgical resection)
* Acute liver disease, unexplained transaminase elevations, or elevated serum calcium
* History of allergic reactions attributed to compounds of similar chemical composition to the study agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Concomitant corticosteroids or anticoagulants needed on a regular or predictable intermittent basis
* New diagnosis of invasive carcinoma
* Use of non-study investigational agent(s) =< 3 months prior to randomization
* Chemotherapy =< 6 months prior to randomization (Note: topical chemotherapy will be assessed on a case-by-case basis)
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Regular use of NSAIDs =< 6 weeks prior to randomization, defined as a frequency of 7 consecutive days (1 week) for > 3 weeks (Exception: low dose aspirin [81 mg] for those subjects who are chronic users of aspirin prior to the beginning of the study)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-08-20 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Sinicrope, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Illinois College of Medicine - Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Acetylsalicylic Acid and Eflornithine): Patients receive 325 mg acetylsalicylic acid PO once daily and 500 mg eflornithine PO once daily on days 1-28.
- Arm II (Placebo): Patients receive corresponding placebo PO daily on days 1-28.
Period: Overall Study
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Started | 54 | 53
Completed | 49 | 49
Not Completed | 5 | 4
Not completed — Cancel Prior to treatment | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Ineligible | 3 | 0

BASELINE CHARACTERISTICS:
Population: All eligible patients that began protocol treatment were included in this analysis. Patients who cancelled prior to treatment, violations and ineligible patients were excluded.
Groups:
- Arm I (Acetylsalicylic Acid and Eflornithine): Patients receive 325 mg acetylsalicylic acid PO once daily and 500 mg eflornithine PO daily on days 1-28.
- Total: Total of all reporting groups
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 83] | 62 [50 to 79] | 62 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 23 | 30 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Recurrence Rate for the Treatment Arm Relative to Placebo
Description: The primary endpoint is the proportion of participants with an adenoma recurrence at the 1-year follow-up colonoscopy exam. All eligible, randomized participants who have signed a consent form and received at least one follow-up endoscopy exam will be considered evaluable for the primary endpoint. This adenoma recurrence rate for DFMO + aspirin will be compared to double placebo to see if there is improvement in the adenoma recurrence rate in this patient population. A 1-sided Chi-square test was used to determine if there was a significant difference between treatment arms.
Time Frame: At 1 year
Population: On Arm 1, 1 patient cancelled prior to treatment, 1 was a violation, 3 were deemed ineligible, and 7 patients did not receive a follow-up endoscopy. On Arm 2, 3 patients cancelled prior to treatment, 1 was a violation, and 6 did not receive a follow-up endoscopy.
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Number analyzed (Participants) | 42 | 43
proportion of participants | 0.595 | 0.581
Statistical Analysis 1: Comparison: Arm I (Acetylsalicylic Acid and Eflornithine) vs Arm II (Placebo); Test type: Superiority; p = 0.448, Chi-squared

2. Secondary Outcome: ACF Characteristics vs Adenoma Recurrence Rate
Description: A potential surrogate endpoint biomarker is the aberrant crypt focus (ACF). ACF are the earliest lesions that can be detected in colorectal mucosa and are believed to be precursors of adenomas and cancers. At the 1-year time point, the presence of adenoma recurrence and the number of ACF sites was recorded for each patient. The percent change in ACF number was calculated as the number of ACF present at the 1-year post-intervention exam minus the baseline number of ACF, divided by the number of ACF present at baseline. A negative score represents a loss in the number of sites and a positive number indicates an increase in the number of ACF sites. Therefore, the possible range in percent change cannot be lower than -100% and has no upper bound. A Wilcoxon Rank-sum test was used to assess the relationship between ACF percent change and adenoma recurrence rate. This analysis was only conducted in those participants who had at least 5 rectal ACF at baseline.
Time Frame: At baseline and 1 year
Population: All patients that were eligible, treated, analyzed for ACF at baseline and 12-months, and had 5 or more ACF at baseline were included in this analysis.
Measure: Median (Full Range); unit: percentage of change in ACF number
Groups:
- All Patients: Patients from Arm I and Arm II were combined in this analysis
Arm/Group | All Patients
Number analyzed (Participants) | 62
percentage of change in ACF number
  No Adenoma Recurrence at 12 months: number analyzed (Participants) | 25
  No Adenoma Recurrence at 12 months | -20.8 [-89.5 to 237.5]
  Adenoma Recurrence at 12 months: number analyzed (Participants) | 37
  Adenoma Recurrence at 12 months | -45.0 [-100 to 300]
Statistical Analysis 1: Comparison: All Patients; This statistical analysis compares the difference between the number of patients with No adenoma recurrence at 12 months with those with adenoma recurrence at 12 months; Test type: Superiority; p = 0.358, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Characterization of ACF
Description: A potential surrogate endpoint biomarker is the aberrant crypt focus (ACF). ACF are the earliest lesions that can be detected in colorectal mucosa and are believed to be precursors of adenomas and cancers. The number and total size of ACF sites may serve as risk markers for adenoma/carcinoma development. The median number of ACF sites per patient were collected prior to treatment.
Time Frame: Baseline
Population: Of the 49 eligible patients receiving treatment in Arm I, 2 patients did not have ACF analysis done. The same number of patients of patients did not have ACF done in Arm II.
Measure: Median (Full Range); unit: number of ACF sites
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Number analyzed (Participants) | 47 | 47
number of ACF sites | 11 [0 to 42] | 7 [0 to 31]

4. Secondary Outcome: Comparison of the Percent Change in ACF Number Across the 2 Treatment Arms
Description: The number of ACF sites per patient was collected at baseline and at 1-year time points. The percent change in ACF number was calculated as the number of ACF present at the 12-month post-intervention exam minus the baseline number of ACF, divided by the number of ACF present at baseline. A negative score represents a loss in the number of sites from baseline to year 1 post-treatment. A positive number indicates an increase in the number of ACF sites. Therefore, the possible range in percent change cannot be lower than -100% and has no upper bound. The percent change in ACF number between arms was compared using a t-test.
Time Frame: At baseline and 12 months
Population: All eligible treated patients that were assessed for ACF at baseline and after 1-year of treatment were included in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of change in ACF number
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Number analyzed (Participants) | 31 | 31
percentage of change in ACF number | -28.6 (51.1) | 10.6 (97.4)
Statistical Analysis 1: Comparison: Arm I (Acetylsalicylic Acid and Eflornithine) vs Arm II (Placebo); Test type: Superiority; p = 0.513, t-test, 2 sided

5. Secondary Outcome: Safety, Tolerability, and Adverse Events of Study Treatment
Description: The National Cancer Institute (NCI) Common Terminology Criteria (CTC) Version 3.0 was used to grade all adverse events. The number of patients reporting a grade 3 or higher event are tabulated here. A grade 3 event is one categorized as being severe or medically significant but not immediately life-threatening. A grade 4 is considered life-threatening, and a grade 5 is death related to the event. A complete list of all adverse events is given in the Adverse Events section.
Time Frame: Up to 48 months from beginning treatment.
Population: On Arm 1, 1 patient cancelled prior to treatment, 1 was a violation, 3 were deemed ineligible. On Arm 2, 3 were ineligible, 1 was a violation. All other patients were treated and evaluated for toxicity and included in this evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Number analyzed (Participants) | 49 | 49
Participants
  Grade 3 Adverse Event | 0 | 3
  Grade 4 Adverse Event | 0 | 0

6. Other Pre Specified Outcome: Effect of the Study Drugs and Placebo With Respect to Biomarkers
Description: For continuous variables, we will use the 2-sample t-test (or nonparametric equivalent) to compare the active arm to the placebo arm. For categorical data, we will explore the relationship between the treatment arms and biomarkers with chi-square or fisher's exact tests. Correlations will be sought between caspase-3 staining, proliferative indices and their ratio, as well as other biomarkers using a chi-square test.
Time Frame: Baseline and 12 months
Population: Data were not collected for this endpoint.
Arm/Group | All Patients
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Gene Expression Analysis
Description: Differences in log-transformed values among ACF or patient characteristics will be compared using t tests or analysis of variance (ANOVAs).
Time Frame: Baseline and 12 months
Population: Data were not collected for this endpoint.
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were collected at the end of each 28 day cycle, for up to 1 year. All patients that received treatment and were assessed for adverse events are included in this section of the report. There was 1 patient cancel and 1 patient not evaluated for adverse events, leaving 52 patients. In Arm 2, there were 3 cancels which left 50 patients evaluated for adverse events.
Arm/Group | Arm I (Acetylsalicylic Acid and Eflornithine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/50
Other Adverse Events (participants affected / at risk) | 4/52 | 4/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Acetylsalicylic Acid and Eflornithine) (N=52) | Arm II (Placebo) (N=50)
Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Acetylsalicylic Acid and Eflornithine) (N=52) | Arm II (Placebo) (N=50)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (7) | 4 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less